CLINICAL TRIAL: NCT05106413
Title: Evaluation of the Clinical Benefit of a Transmitter for Contralateral Routing of Signals (CROS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This clinical trial has been early terminated due to recruiting issues of the calculated sample size.
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-377
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2021-11

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech Intelligibility with CROS device (Experimental): The focus of this study is on Speech Intelligibility (SI), evaluated by the Oldenburg Sentence test (OLSA), which measures a speech recognition threshold (SRT) in dB SNR (signal to noise ratio).
  Therefore each participant will perform the tests with the experimental rechargeable CROS transmitter (CROS) in different interventions, like comparison to monaural fitting and unaided condition.
  All participants will perform the same tests. The order of the intervention in the speech test is randomized, but will be performed in the same visit by each participant.
  Interventions: Other: BiCROS fitting; Other: Monaural fitting; Other: Unaided condition; Other: CROS baseline

INTERVENTIONS:
Other: BiCROS fitting — Each participant will be fitted with the experimental CROS device on the poorer, unaidable ear and with a compatible hearing device on the other ear.
Other: Monaural fitting — Each participant will be fitted with a hearing aid on the better hearing ear and no device on the poorer, unaidable ear.
  Monaural hearing aid fitting acts as control intervention.
Other: Unaided condition — No treatment, i.e. the participants are not fitted with a CROS device and/ or hearing aid.
  Unaided condition acts as control intervention.
Other: CROS baseline — Each participant will be fitted with the experimental CROS device on the poorer, unaidable ear and with a compatible device on the other ear. The difference to the BiCROS condition is the setup of the microphones in the CROS device and the compatible hearing device.
  This test condition is only tested for speech intelligibility in diffuse noise and acts as control intervention.

SUMMARY:
This study will evaluate the clinical benefit of a transmitter for contralateral routing of signals. The benefit will be evaluated in noisy environments regarding speech intelligibility when the CROS system is adjusted to different microphone settings. Additionally, data regarding overall system stability, crash reboot rate, sound quality and connectivity will be obtained over a period of time to validate the CROS system in combination with smartphone and accessories. This study is a confirmatory study.

DETAILED DESCRIPTION:
Unilateral Hearing Loss (UHL) can be defined as any degree of permanent hearing loss on one ear with normal hearing in the opposite ear. Unilateral hearing loss can be debilitating associated with audiological, psychosocial and educational challenges. Audiological challenges include the reduced ability to localize sounds, reduced awareness on the unaidable side and difficulties hearing in noise or at a distance.

One solution for unaidable UHL is Contralateral Routing of Signals (CROS) and Bilateral Contralateral routing of signals (BiCROS) using a so- called CROS transmitter together with a hearing aid.

The rationale for this clinical investigation is to collect clinical data with a rechargeable CROS transmitter to evaluate the benefits of a BiCROS fitting compared to the alternative treatment option, the monaural hearing aid fitting, and to no treatment in noisy listening situations.

ELIGIBILITY:
Inclusion Criteria:

* hearing impaired adults, with & w/o hearing aids (experiences)
* good written and spoken (Swiss) German language skills
* ability to fill in a questionnaire conscientiously
* informed consent as documented by signature
* asymmetric hearing loss: one unaidable ear (min. N6 hearing loss) / the other ear with N3 or N4 hearing loss
* availability of Smartphone
* availability of TV or Tablet
* ability to operate and handle the investigational device
* ability to describe listening impressions/experiences and the use of the hearing aid
* Ability to produce a reliable hearing test result

Exclusion Criteria:

* Contraindications to the medical device:
* aidable hearing loss on the intended CROS side
* acute tinnitus (in either one ear and occurrence less than three months)
* anatomical deformity of the CROS ear (e.g. absence of the auricle)
* Known hypersensitivity or allergy to materials of the investigational device
* any auricle deformities, that prevents secure placement of the (test) devices
* no willingness to test the investigational device system
* no willingness to test the investigational device system for at least 8h a day
* Hint for psychological problems from investigators point of view
* reported fluctuating hearing that could influence the test result
* reported symptoms of vertigo and dizziness by participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Speech Intelligibility (SI) in noise (fix direction): BiCROS fitting vs. monaural hearing aid fitting | 2 weeks
  The primary objective of this clinical investigation is to evaluate whether a BiCROS fitting (better ear fitted with a hearing device, unaidable ear supplied with a CROS device) improves speech intelligibility in noise compared to a monaural fitting (just the aidable ear is supplied by a hearing aid), for adults with an asymmetric hearing loss, measured with the Oldenburg Sentence Test (OLSA). Results of the speech test will be the SRT (speech recognition threshold) in dB SNR (signal to noise ratio).
  The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).

SECONDARY OUTCOMES:
SI in noise (fix direction): BiCROS fitting vs. unaided | 2 week
  A secondary objective of this clinical investigation is to evaluate whether a BiCROS fitting improves speech intelligibility in noise compared to an unaided condition, for adults with an asymmetric hearing loss, measured with the Oldenburg Sentence Test (OLSA).
  Results of the speech test will be the SRT (dB SNR). The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SI in diffuse noise: BiCROS fitting vs. monaural fitting | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a BiCROS fitting improves speech intelligibility by at least 1 dB SNR for 50% SRT in diffuse noise, compared to a monaural hearing aid fitting.
  The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SI in diffuse noise: BiCROS fitting vs. unaided | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a BiCROS fitting improves speech intelligibility by at least 1 dB SNR for 50% SRT in diffuse noise, compared to an unaided condition.
  The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SI in diffuse noise: BiCROS vs. CROS baseline fitting | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a BiCROS fitting improves speech intelligibility in diffuse noise compared with a CROS baseline fitting. CROS baseline means a fitting of an additional program with different hearing instrument microphone setup.
  The SI will be tested with the OLSA in diffuse noise. The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SI in diffuse noise: CROS baseline fitting vs. unaided | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a CROS baseline fitting improves speech intelligibility in diffuse noise compared with an unaided condition.
  The SI will be tested with the OLSA in diffuse noise. The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SI in diffuse noise: CROS baseline fitting vs. monaural fitting | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a CROS baseline fitting improves speech intelligibility in diffuse noise compared with a monaural fitting.
  The SI will be tested with the OLSA in diffuse noise. The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
SP in diffuse noise: monaural fitting vs. unaided | 2 weeks
  A secondary objective of this clinical investigation is to evaluate whether a monaural fitting improves speech intelligibility in diffuse noise compared with an unaided condition.
  The SI will be tested with the OLSA in diffuse noise. The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 70 dB (A).
Evaluation of Sound quality | 3 weeks
  A secondary objective of this study is to evaluate the participant's satisfaction of the sound quality of the experimental CROS device by a subjective rating during a three-week home trial period.
  Scale: very unsatisfied- unsatisfied- neither nor- satisfied- very satisfied
Evaluation of System stability | 3 weeks
  A secondary objective of this study is to evaluate the participant's satisfaction of the system stability of the experimental CROS device during a three-week home trial period.
  The participant shall report, if there are artefacts audible: never/ 1-2 times a week/ 3-6 times a week/ daily
Evaluation of streaming | 3 weeks
  A secondary objective of this study is to evaluate the participant's satisfaction of the streaming sound quality of the experimental CROS device, by a subjective rating during a three-week home trial period.
  Scale: very unsatisfied- unsatisfied- neither nor- satisfied- very satisfied
Evaluation of listening effort | 3 weeks
  A secondary objective is to evaluate the subjective listening effort in noise reported by the participant whilst wearing the experimental CROS device.
  Scale: not at all - slightly - somewhat - moderately - very - extremely

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Bagatto M, DesGeorges J, King A, Kitterick P, Laurnagaray D, Lewis D, Roush P, Sladen DP, Tharpe AM. Consensus practice parameter: audiological assessment and management of unilateral hearing loss in children. Int J Audiol. 2019 Dec;58(12):805-815. doi: 10.1080/14992027.2019.1654620. Epub 2019 Sep 5. PMID 31486692
- [Background] Snapp HA, Hoffer ME, Spahr A, Rajguru S. Application of Wireless Contralateral Routing of Signal Technology in Unilateral Cochlear Implant Users with Bilateral Profound Hearing Loss. J Am Acad Audiol. 2019 Jul/Aug;30(7):579-589. doi: 10.3766/jaaa.17121. Epub 2018 Dec 13. PMID 30541657
- [Background] Snapp H. Nonsurgical Management of Single-Sided Deafness: Contralateral Routing of Signal. J Neurol Surg B Skull Base. 2019 Apr;80(2):132-138. doi: 10.1055/s-0039-1677687. Epub 2019 Jan 17. PMID 30931220
- [Background] Lieu JE, Tye-Murray N, Karzon RK, Piccirillo JF. Unilateral hearing loss is associated with worse speech-language scores in children. Pediatrics. 2010 Jun;125(6):e1348-55. doi: 10.1542/peds.2009-2448. Epub 2010 May 10. PMID 20457680
- [Background] McKay S, Gravel JS, Tharpe AM. Amplification considerations for children with minimal or mild bilateral hearing loss and unilateral hearing loss. Trends Amplif. 2008 Mar;12(1):43-54. doi: 10.1177/1084713807313570. PMID 18270178